CLINICAL TRIAL: NCT07173816
Title: Optimizing PrEP Uptake for African American Women in the South by Empowering Women to Make Informed HIV Prevention and Sexual Health Choices
Acronym: EMPOWER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mohammad Rifat Haider, Assistant Professor, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: R34MH137775 (NIH); R34MH137775 (NIH)
Record Dates: First submitted 2025-09-01; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: HIV Pre-exposure Prophylaxis

STUDY DESIGN:
Intervention Model Description: Investigators will recruit 80 Black women from HIV testing sites who have engaged in HIV risk behavior in the prior three months and randomly assign them to either the EMPOWER intervention condition (n=40) or a standard of care control condition (n=40). Standard of care includes provision of opt-out PrEP. Both conditions will receive EMPOWER. However, the standard of care control condition will receive the intervention after the 3-month follow-up assessment. The active intervention period will last 9 weeks (5 weekly sessions and a booster session after 4 weeks).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator): This arm will receive the intervention first.
  Interventions: Behavioral: EMPOWER
- Waitlist Control (Active Comparator): This arm will receve the intervention after the wait period
  Interventions: Behavioral: EMPOWER

INTERVENTIONS:
Behavioral: EMPOWER — EMPOWER, a group-based 6 sessions telehealth behavioral intervention, will comprise sexual health goals and values elicitation, sexual health plan development, and motivational enhancement skills will be used to promote effective HIV prevention decision-making within the relationship context, incorporating the sexual values of each participant. This will allow each participant to develop a personalized, tailored sexual health plan that includes PrEP deliberation to enhance PrEP decision-making, uptake and persistence within a culturally congruent and empowering program that aims to reduce stigma around HIV and barriers to access.

SUMMARY:
Pilot testing of EMPOWER, a group sexual health intervention, to increase uptake and persistence of PrEP

DETAILED DESCRIPTION:
This study will pilot test the telehealth intervention EMPOWER (Enhancing and Motivating PrEP Options among Women through Empowerment and Resilience) by adapting an evidence-informed intervention, POWER (Progressing Our Well-Being, Emotions, and Relationships) based on mindfulness and cognitive behavioral therapy, to improve PrEP uptake and persistence by Black women in the South.

Conduct a waitlist-controlled, randomized pilot trial of the 6-session group intervention using a crossover design with 80 Black women. Clinical outcomes will be the PrEP uptake and PrEP persistence measured by TDF via the dried blood spot at baseline, 3- and 6-months post-intervention. We will also assess the intervention's feasibility, acceptability, and usability. The outcomes will be compared with the usual standard of care (opt-out PrEP) at the intervention site.

ELIGIBILITY:
Inclusion Criteria:

1. Identification as cis-gendered Black woman;
2. Age 18 and older;
3. Engaging in risky sexual behavior in prior 3 months (condomless vaginal or anal sex with a non-main partner, or a partner with known or suspected risk behavior such as injection drug use or HIV/STI, multiple sex partners, transactional sex);
4. Access to a device with a screen, a web browser, and adequate internet speed (e.g., smartphone, computer) for videoconferencing;
5. Able to speak and read English; and
6. No plans to leave the Atlanta, GA area during the duration of study participation.

Exclusion Criteria:

1. Cognitive or mental health condition that limits the ability to provide informed consent;
2. Self-reported use of PrEP or PEP medication in the past three months;
3. Unable to speak and read English; and
4. Currently living with HIV.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women
Enrollment: 80 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of EMPOWER Intervention | From enrollment to the end of data collection and analysis at 6 months
  Enrollment rate will be used an indicator of the feasibility of the intervention
Acceptability of EMPOWER Intervention | From enrollment to the end of data collection and analysis at 6 months
  Acceptability of the intervention based on participant satisfaction using the Client Satisfaction Questionnaire scores

CONTACTS AND LOCATIONS:
Locations (1):
- Empowerment Resource Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
Investigators will not share the IPD of the participants of this study with others because the investigaotrs will only report the aggregated results of the study.